CLINICAL TRIAL: NCT07028320
Title: A Multicenter, Randomized, Open-label, Parallel Controlled, Phase Ⅲ Clinical Study to Evaluate the Efficacy and Safety of SAL056 (Teriparatide for Injection ) in the Treatment of Postmenopausal Women With Osteoporosis at High Fracture Risk
Brief Title: To Evaluate the Efficacy and Safety of SAL056 for Postmenopausal Women With Osteoporosis at High Fracture Risk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAL056A301
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Postmenopausal Women With Osteoporosis
Keywords: Postmenopausal Women With Osteoporosis; Teriparatide
MeSH Terms: interventions — Teriparatide; Injections; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: SAL056 (56.5μg) (Experimental): Administered by subcutaneous injection once a week during treatment phase
  Interventions: Drug: SAL056 (56.5μg)
- Drug: Alendronate (Active Comparator): 70 mg tablet taken once a week during treatment phase
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: SAL056 (56.5μg) — Administered by subcutaneous injection once a week during treatment phase
  Other Names: Teriparatide for Injection
  Arms: Drug: SAL056 (56.5μg)
Drug: Alendronate — 70 mg tablet taken once a week during treatment phase
  Arms: Drug: Alendronate

SUMMARY:
To Evaluate the Efficacy and Safety of SAL056 for Postmenopausal Women with Osteoporosis at High Fracture Risk

DETAILED DESCRIPTION:
The trial consists of a screening period (4 weeks), an open-label treatment period (up to 48 weeks), and a follow-up period (1 weeks), totaling approximately 53 weeks. Subjects who withdraw early will be asked to complete an end of treatment visit, and a safety follow-up visit 2 weeks after the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women with the ability to live independently (≥45 and ≤80 years);
2. The patient has a body mass index(BMI) of 18.0 kg/m2 to 30 kg/m2； The patient has one of the following diagnostic criteria for osteoporosis and subject has at least 2 consecutive vertebrae region (L1 to L4) that are evaluable by dual-energy x-ray absorptiometry (DXA)，a) History of hip/vertebra fragility fracture and bone mineral density (BMD) T-score ≤-1; b）the axial bone (lumbar , femoral neck or total hip) mineral density (BMD) T-score ≤-2.50;c) Bone mineral density (BMD) T-score ≥-2.5 and ≤-1 with proximal humerus, pelvis, or distal forearm end fragility fracture

Exclusion Criteria:

1. In addition to postmenopausal osteoporosis, the other diseases affecting bone metabolism;
2. Patients with other diseases affecting calcium or bone metabolism;
3. Received anti-osteoporosis treatment that does not meet protocol requirements;
4. Received medication that affects bone metabolism prior to screening, or is planned to use prohibited drugs/non-drug therapy under the protocol during the study period;
5. Patients requiring long-term or continuous use of digoxin and other digitalis drugs during the trial;
6. Patients with other severe underlying diseases； Patients with abnormal indicators that does not meet protocol requirements during the screening periodlaboratory tests

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 493 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) of Lumbar Spine from Baseline to 48 Weeks | Baseline to 48 Weeks
  Percent Change in Bone Mineral Density (BMD) of Lumbar Spine from Baseline to 48 Weeks

SECONDARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) of Lumbar Spine from Baseline to 24 Weeks | Baseline to 24 Weeks
  Percent Change in Bone Mineral Density (BMD) of Lumbar Spine From Baseline to 24 Weeks
Percent Change in Bone Mineral Density (BMD) of Total Hip from Baseline to 24/48 Weeks | Baseline to 24/48 Weeks
  Percent Change in Bone Mineral Density (BMD) of Total Hip From Baseline to 24/48 Weeks
Percent Change in S-CTX and P1NP From Baseline to12/ 24/48 Weeks | Baseline to 12/24/48 Weeks
  Percent Change in S-CTX and P1NP From Baseline to 12/24/48 Weeks
Proportion of Subjects with New Fragility Fractures from Baseline to 24/48 Week | Baseline to 24/48 Weeks
  Proportion of Subjects With New Fragility Fractures from Baseline to 24/48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Lin Zhang, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hosptital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No